CLINICAL TRIAL: NCT02296190
Title: Multi-Center, Placebo-Controlled, Dose-Ranging Phase 2 Electrophysiological Study of Intranasal Administration of MSP-2017 for the Conversion of Induced Paroxysmal Supraventricular Tachycardia (PSVT) to Sinus Rhythm
Brief Title: Efficacy and Safety of Intranasal MSP-2017 (Etripamil) for the Conversion of PSVT to Sinus Rhythm
Acronym: NODE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milestone Pharmaceuticals Inc. (Other)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSP-2017-1109
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Results first posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Paroxysmal Supraventricular Tachycardia (PSVT)
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — etripamil

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: If, during the double-blind study, PSVT could not be induced, the mechanism of PSVT was neither atrioventricular (AV) reentrant tachycardia (AVRT) nor AV nodal reentrant tachycardia (AVNRT), or it was not possible to sustain an episode of PSVT for 5 minutes in a subject who previously provided written informed consent for substudy participation, the subject was eligible to participate in the optional open-label substudy.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etripamil (Experimental): 1 dose of Etripamil via 4 intranasal applications at time 0 (140 mg, 105 mg, 70 mg, or 35 mg)
  Interventions: Drug: Etripamil
- Placebo (Placebo Comparator): 1 dose of placebo via 4 intranasal applications at time 0
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etripamil — intranasal administration via 4 prefilled Aptar Pharma Unit-Dose Spray devices
  Other Names: MSP-2017
  Arms: Etripamil
Drug: Placebo — intranasal administration via 4 prefilled Aptar Pharma Unit-Dose Spray devices
  Arms: Placebo

SUMMARY:
The primary objective of this study is to demonstrate the superiority of at least 1 dose of intranasal (IN) MSP-2017 (Etripamil) over placebo in terminating PSVT induced in an electrophysiology (EP) laboratory.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, dose-ranging study to evaluate the effects of 4 different doses of MSP-2017 (Etripamil) in subjects with paroxysmal supraventricular tachycardia. It includes an up to 21-day Screening Period, a 1-day Treatment Visit, and either a Follow-up Visit or Early Termination Visit occurring 12 hours to 5 days after the Treatment Visit. Subjects will be randomized to yield at least 100 evaluable subjects distributed into 5 groups of at least 20 subjects each.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years and older at Screening
* Has a history of PSVT
* Is scheduled for an electrophysiology study and catheter ablation
* Has provided written informed consent
* Agrees to use a medically accepted form of contraception or abstinence to prevent pregnancy. Males must agree to use an acceptable form of contraception or abstinence from the time of study drug administration through the Follow-up Visit. Females must agree to use an acceptable form of contraception or abstinence from Screening until 30 days following study drug administration. Post-menopausal female subjects must be amenorrheic for ≥ 12 months prior to Screening or ≥ 6 weeks post-surgical bilateral oophorectomy (with or without hysterectomy) prior to Screening, if they do not wish to use an acceptable form of contraception or abstinence. Acceptable forms of contraception include: A condom and an intrauterine device; A condom and hormonal contraception; A condom and a diaphragm; Sterilization of the subject or the subject's partner(s) (sterilization procedure must have been performed 3 or more months prior); Hysterectomy of the subject or the subject's partner(s)
* If a female of childbearing potential: Has a negative serum pregnancy test result at Screening (Screening must occur ≥7 days prior to randomization [ie, on or before Day -7]) and at the Treatment Visit (pre-PSVT induction); Has had a menstrual period within 28 days of the Treatment Visit.

Exclusion Criteria:

* Has a history of serious allergic reaction to verapamil (especially when administered intravenously) including rash, itching or swelling (especially of the face, tongue, or throat), severe dizziness, or trouble breathing
* Is currently participating in another drug or device study, or has received an investigational drug or device within 30 days of Screening
* Has evidence of clinically significant cardiovascular, endocrine, gastrointestinal, hematologic, hepatic, immunologic, neurologic, oncologic, pulmonary, psychiatric, or renal disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of study results
* Is a female who is breast feeding, pregnant, or planning to become pregnant during the study period
* Has evidence of any clinically significant acute or chronic condition of the nasal cavity (e.g., rhinitis or deviated septum) which could interfere with IN administration of the study drug in either or both nasal cavities
* Has any of the following at screening or at the Treatment Visit: Systolic blood pressure <100 mmHg, Diastolic blood pressure <50 mmHg
* Has evidence of hepatic impairment, defined as: Alanine aminotransferase or aspartate aminotransferase levels that are greater than or equal to 3× upper limit of normal (ULN) or Bilirubin levels that are greater than or equal to 2× ULN, unless due to Gilbert's syndrome
* Has evidence of renal impairment, defined as an estimated glomerular filtration rate <30 mL/min (Modification of Diet in Renal Disease method)
* Has taken digoxin, verapamil, diltiazem, or any Class I, II (e.g., beta blockers), or III antiarrhythmic drug less than the equivalent of 5 half-lives of this drug prior to the Treatment Visit
* Has taken amiodarone within 30 days of the Treatment Visit
* Has taken drugs of abuse which, in the opinion of the Investigator, would impact the validity of study results
* Has had myocardial infarction, percutaneous coronary intervention, cerebrovascular accident, transient ischemic attack, unstable angina, or acute decompensation of heart failure within 6 months of Screening
* Has a history or evidence of second- or third-degree atrioventricular block
* Has an implanted device (e.g., pacemaker, or implantable cardioverter defibrillator) that precludes study participation in the opinion of the Investigator and Study Medical Monitor
* Has a history or evidence of preexcitation syndrome (e.g., Wolff-Parkinson- White syndrome, short PR, etc.)
* Has evidence of a QT interval (Bazett's correction) (QTcB) >455 milliseconds at Screening or at the Treatment Visit
* Has a history or evidence of familial long QT syndrome, torsades de pointes, ventricular fibrillation, sustained ventricular tachycardia, Brugada syndrome, or sudden cardiac death
* Has evidence of recurrent or chronic atrial tachycardia, atrial flutter, or atrial fibrillation; that could interfere with the current investigation; or
* Has a history or evidence of congestive heart failure (except New York Heart Association Class I) or pulmonary edema

In addition, randomized subjects who meet any of the following criteria at the Treatment Visit (Day 1) prior to study drug administration, will be excluded from participation in the study:

* PSVT cannot be induced or the mechanism of PSVT is neither Atrioventricular reentrant tachycardia (AVRT) nor Atrioventricular nodal reentry tachycardia (AVNRT)
* It is not possible to sustain an episode of PSVT for 5 minutes
* The subject requires a continuous sedative (e.g., propofol), continuous analgesic, or inhaled anesthetic at any point until time 30. Minimally necessary dose(s) of benzodiazepine(s) (e.g., midazolam) and/or narcotic(s) (e.g., fentanyl) (given via single or multiple administration[s]) may be used at the Investigator's discretion. The identity(-ies) and actual administered dose(s) of any benzodiazepine(s) and/or narcotic(s) should be recorded in the study documentation. Local anesthetic(s) may be used at the Investigator's discretion; any use should be recorded in the study documentation
* The subject has undergone prior ablation, and the subject's atrioventricular node function is abnormal in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2015-03-27; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Plat, Study Director — Chief Medical Officer
Locations (30):
- United States (26):
  - Arizona Heart Rhythm Center, Phoenix, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mercy General Hospital, Sacramento, California
  - South Denver Cardiology Associates, Littleton, Colorado
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Northside Hospital, St. Petersburg, Florida
  - University of South Florida Health South Tampa Center, Tampa, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Iowa Heart Center, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - MedStar Health Research Institute, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Aultman Hospital Cardiology Clinical Trials, Canton, Ohio
  - University of Cincinnati Medical Center Division of Cardiovascular Diseases, Cincinnati, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Great Lakes Medical Research, LLC, Willoughby, Ohio
  - Black Hills Cardiovascular Research, Rapid City, South Dakota
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Baylor St. Luke's Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Centra Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Canada (4):
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - The Montreal Heart Institute, Montreal, Quebec
  - CHUM Hotel Dieu, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stambler BS, Dorian P, Sager PT, Wight D, Douville P, Potvin D, Shamszad P, Haberman RJ, Kuk RS, Lakkireddy DR, Teixeira JM, Bilchick KC, Damle RS, Bernstein RC, Lam WW, O'Neill G, Noseworthy PA, Venkatachalam KL, Coutu B, Mondesert B, Plat F. Etripamil Nasal Spray for Rapid Conversion of Supraventricular Tachycardia to Sinus Rhythm. J Am Coll Cardiol. 2018 Jul 31;72(5):489-497. doi: 10.1016/j.jacc.2018.04.082. PMID 30049309

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults aged 18 years and older with Paroxysmal supraventricular tachycardia (PSVT) who met the study inclusion/exclusion criteria. Study was initiated on March 27, 2015 and completed on December 8, 2016 and was performed in electro-physiology clinics in the USA and Canada.
Groups:
- Etripamil_140 mg; Etripamil_ 105 mg; Etripamil_70 mg; Etripamil_35 mg: 1 dose of Etripamil via 4 prefilled Aptar Pharma Unit-Dose Nasal Spray devices.
- Placebo: 1 dose of Placebo via 4 prefilled Aptar Pharma Unit-Dose Nasal Spray devices.
- Open-label Etripamil 70 mg: 9 subjects were assigned to an open-label Sub-study Safety Population. Subjects participating in the open-label sub-study received intra nasal administration of 70 mg MSP-2017 (total) via 2 prefilled Aptar Pharma Unit-Dose Spray devices.
Period: Overall Study
Arm/Group | Etripamil_140 mg | Etripamil_ 105 mg | Etripamil_70 mg | Etripamil_35 mg | Placebo | Open-label Etripamil 70 mg
Started | 35 | 41 | 35 | 43 | 36 | 9
Completed | 21 | 20 | 23 | 20 | 20 | 9
Not Completed | 14 | 21 | 12 | 23 | 16 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Failure to induce PSVT | 6 | 10 | 5 | 13 | 8 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — PSVT < 5 minutes | 5 | 6 | 6 | 6 | 5 | 0
Not completed — Patient was given Propofol | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Patient with Atrial Tachycardia | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Blood pressure <100 after sedation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Atrial Tachycardia induced not PSVT | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Patient on antiarrhythmic medication | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Failed PSVT with mechanism of AVNRT | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lab result not available in time | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (all randomized participants who received at least 1 dose of study drug)
Groups:
- Etripamil_105 mg; Etripamil_70 mg; Etripamil_35 mg; Open- Label Etripamil 70 mg: 1 dose of Etripamil via 4 prefilled Aptar Pharma Unit-Dose Nasal Spray devices.
- Total: Total of all reporting groups
Arm/Group | Etripamil_140 mg | Etripamil_105 mg | Etripamil_70 mg | Etripamil_35 mg | Placebo | Open- Label Etripamil 70 mg | Total
Number analyzed (Participants) | 21 | 20 | 23 | 20 | 20 | 9 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 17 | 19 | 19 | 18 | 9 | 96
  >=65 years | 7 | 3 | 4 | 1 | 2 | 0 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 9 | 14 | 10 | 6 | 65
  Male | 8 | 7 | 14 | 6 | 10 | 3 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 17 | 14 | 18 | 17 | 18 | 7 | 91
  BLACK OR AFRICAN AMERICAN | 2 | 4 | 3 | 2 | 2 | 1 | 14
  OTHER | 2 | 2 | 2 | 0 | 0 | 1 | 7
  ASIAN | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 7 | 4 | 7 | 4 | 0 | 26
  United States | 17 | 13 | 19 | 13 | 16 | 9 | 78

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Successfully Converted From PSVT to Sinus Rhythm Within 15 Minutes of Study Drug Administration
Description: The primary efﬁcacy endpoint was the rate of successful PSVT conversion to sinus rhythm lasting at least 30 seconds within 15 minutes of study drug administration after a minimum of 5 minutes in sustained PSVT.
Time Frame: Within 15 minutes of study drug administration
Population: The efficacy analysis was based on the Evaluable Population which included all randomized subjects who were induced and sustained Supraventricular tachycardia (SVT) for 5 minutes, received the study drug, and completed the assessment of conversion to sinus rhythm.
  The "Open- Label Etripamil 70 mg" group was not part of the Evaluable Population, as the subjects did not meet the criteria of having sustained Supraventricular tachycardia (SVT) for 5 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Etripamil_140 mg | Etripamil_ 105 mg | Etripamil_70 mg | Etripamil_35 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 23 | 20 | 20
Participants | 20 | 15 | 20 | 13 | 7
Statistical Analysis 1: Comparison: Etripamil_140 mg vs Etripamil_ 105 mg vs Etripamil_70 mg vs Etripamil_35 mg vs Placebo; Statistical analysis was performed with the Fisher's exact test to compare the conversion rate between the MSP-2017 groups and the placebo group; Test type: Superiority; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time of study drug administration (Treatment Visit Day 1) until study participation completed at the Follow-up Visit which occurred from 12 hours to up to 5 days after the Treatment Visit. Maximum time frame 6 days.
Groups:
- Open Label Etripamil 70 mg: 1 dose of Etripamil via 4 prefilled Aptar Pharma Unit-Dose Nasal Spray devices.
Arm/Group | Etripamil_140 mg | Etripamil_105 mg | Etripamil_70 mg | Etripamil_35 mg | Placebo | Open Label Etripamil 70 mg
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/23 | 0/20 | 0/20 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/21 | 3/20 | 0/23 | 0/20 | 1/20 | 0/9
Other Adverse Events (participants affected / at risk) | 20/21 | 14/20 | 18/23 | 17/20 | 4/20 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etripamil_140 mg (N=21) | Etripamil_105 mg (N=20) | Etripamil_70 mg (N=23) | Etripamil_35 mg (N=20) | Placebo (N=20) | Open Label Etripamil 70 mg (N=9)
Bundle Branch Block Right (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etripamil_140 mg (N=21) | Etripamil_105 mg (N=20) | Etripamil_70 mg (N=23) | Etripamil_35 mg (N=20) | Placebo (N=20) | Open Label Etripamil 70 mg (N=9)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7) | 11 (11) | 12 (12) | 1 (1) | 6 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 9 (9) | 6 (6) | 5 (5) | 0 (0) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4) | 7 (7) | 5 (5) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Increased lacrimation (Eye disorders) | 5 (5) | 1 (1) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Atrioventricular block second-degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7) | 8 (8) | 9 (9) | 2 (2) | 1 (1)
Upper -Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enlarged uvula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palatal Swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle Branch Block Right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter Site Haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular complication associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurogenic Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular Block Complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post Procedural Complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes